CLINICAL TRIAL: NCT02785991
Title: Prospective Observational Study of Pulmonary Vein Cryoablation in Subjects With Atrial Fibrillation (AF) in Spain
Brief Title: Spanish Registry of Cryoballoon Ablation
Acronym: RECABA
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: RECABA
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Balloon cryoablation — pulmonary vein cryoablation for atrial fibrillation

SUMMARY:
The purpose of this registry is to reflect on standard clinical practice in pulmonary vein cryoablation in Spanish hospitals, the different procedure protocols, details of intervention, complications, long-term follow-up strategy and results in these subjects.

DETAILED DESCRIPTION:
With this study the investigators propose the performance of a prospective registry of pulmonary vein cryoablation in subjects with paroxysmal or persistent AF at Spanish sites to estimate evaluate the efficacy of the cryoablation procedure at 12 months, defined as the absence of recurrences of atrial fibrillation.

Secondary objectives are also defined as:

* Description of the profile of subjects who undergo this type of procedure (demographic factors, cardiovascular risk factors, medication, physical activity, sleep apnea, alcohol, smoking, chronic pulmonary disease, obesity, etc.).
* To evaluate the acute efficacy of the procedure: complete isolation of the pulmonary veins demonstrated by the successful electrical disconnection of the pulmonary veins in the cryoablation procedure.
* Description of the complications related to the procedure.
* To evaluate the use of healthcare resources which this cryoablation procedure entails.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the Data Release Form
* Subjects ≥ 18 years old
* Subjects who meet the indication for the Cryoballoon Ablation procedure.

Exclusion Criteria:

* Subjects with a life expectancy of less than 12 months.
* Subjects who meet the exclusion criteria defined by local legislation (e.g., age, pregnancy, breastfeeding, etc.).
* Subjects who may currently be enrolled, or who plan to take part, in a study with a drug or device that may cause bias during the course of this study.
* Co-participation in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size will be approximately 1000 subjects who must be enrolled over the two-year period, based on the annual rate of cryoballoon ablations carried out in Spain.
Sampling Method: Probability Sample
Enrollment: 1742 (Actual)
Dates: Start 2016-07; Primary Completion 2020-04 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Daniel Martínez Alday, MD, Principal Investigator — Hospital de Basurto; Ermengol Vallés, MD, Principal Investigator — Hospital del Mar; Rocío Cozar, MD, Principal Investigator — Hospital Virgen del Rocío; Angel Ferrero, MD, Principal Investigator — Hospital Clínico de Valencia; Arcadio García Alberola, MD, Principal Investigator — Hospital Virgen de la Arrixaca
Locations (28):
- Spain (28):
  - Hospital Trias i Pujol, Badalona, Barcelona
  - H. Josep Trueta, Girona, Barcelona
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Araba, Alava
  - Hospital Clínico Univeristario San Juan de Alicante, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Clinica Zorrotzaurre, Bilbao
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Reína Sofía, Córdoba
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - H. Universitario Insular de las Palmas, Las Palmas de Gran Canaria
  - Fundación Jiménez Díaz, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - H. C. U. Virgen de la Victoria, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Nisa-Aljarafe, Seville
  - Hospital Virgen Macarena, Seville
  - H.General de Valencia, Valencia
  - Hospital Quirón Salud Valencia, Valencia
  - Hospital Universitario Clínico de Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol

REFERENCES:
- [Derived] Alvarez-Ortega CA, Solorzano Guillen CR, Barrera Cordero A, Toquero Ramos JE, Martinez-Alday JD, Grande Morales CE, Rodriguez Gonzalez A, Garcia Alberola A, Perez Alvarez L, Ferrero de Loma Osorio A, Hernandez Afonso JS, Cozar Leon R, Cano Perez O, Trucco E, Peinado Peinado R. Repeat cryoablation as a redo procedure for atrial fibrillation ablation: Is it a good choice? Cardiol J. 2024;31(2):193-204. doi: 10.5603/CJ.a2023.0017. Epub 2023 Mar 13. PMID 36908163
- [Derived] Ferrero-De-Loma-Osorio A, Cozar R, Garcia-Alberola A, Valles E, Barrera A, Toquero J, Ormaetxe JM, Sanchez JM, Ruiz-Granell R, Amador PB, Rubio JM, Marti-Amor J, Pascual P, Molina I, Martinez-Alday JD; RECABA Investigators. Primary results of the Spanish Cryoballoon Ablation Registry: acute and long-term outcomes of the RECABA study. Sci Rep. 2021 Aug 26;11(1):17268. doi: 10.1038/s41598-021-96655-3. PMID 34446764

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Atrial Fibrillation: Patients With Atrial Fibrillation who meet the indication, according to current clinical practice guidelines, for the Balloon Cryoablation procedure.
Period: Overall Study
Arm/Group | Patients With Atrial Fibrillation
Started | 1742
Completed | 1741
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With Atrial Fibrillation: Patients with paroxysmal and persistent atrial fibrillation who meet criteria to receive a cryoablation procedure.
Arm/Group | Patients With Atrial Fibrillation
Number analyzed (Participants) | 1742
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 543
  Male | 1199
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data not collected
Region of Enrollment [Number; unit: participants]
  Spain | 1742
Demographic factors, cardiovascular risk factors (arterial hypertension, diabetes mellitus, dyslipid [Number; unit: percentage of patients]
  Hypertension | 46.3
  Dyslipidemia | 34.7
  Diabetes Mellitus | 9.1
  Smokers | 13.3
  Ischemia Stroke/TIA | 5.3

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of the Cryoablation Procedure at 12 Months, Defined as the Absence of Recurrences of Atrial Fibrillation.
Description: Percentage of patients freedom from Recurrences of Atrial Fibrillation at 12 months (on ECG, Holter monitor with a duration of at least 30 seconds or implantable devices or event recording systems).
Time Frame: 12 months
Measure: Number; unit: percentage of patients freedom from AF
Groups:
- Patients With Atrial Fibrillation: Patients with paroxysmal and persistent atrial fibrillation
Arm/Group | Patients With Atrial Fibrillation
Number analyzed (Participants) | 1628
percentage of patients freedom from AF | 79

2. Secondary Outcome: The Acute Efficacy of the Procedure:
Description: Complete isolation of the pulmonary veins demonstrated by the successful electrical disconnection of the pulmonary veins in the cryoablation procedure.
Time Frame: 24-48h
Measure: Number; unit: participants
Groups:
- Patients With Paroxysmal and Persistent Atrial Fibrillation: Patients with AF paroxysmal or persistent who meet the criteria for a cryoablation of pulmonary veins.
Arm/Group | Patients With Paroxysmal and Persistent Atrial Fibrillation
Number analyzed (Participants) | 1741
participants | 1726

3. Secondary Outcome: Number of Adverse Events Related to the Procedure
Description: The outcome measure is the number of Adverse Events Related to the Procedure
Time Frame: Up 30 days post procedure
Measure: Number; unit: adverse events
Arm/Group | Patients With Paroxysmal and Persistent Atrial Fibrillation
Number analyzed (Participants) | 1741
adverse events | 120

ADVERSE EVENTS:
Time Frame: Adverse events were collected during enrollment and follow up phase, 32 months.
Description: A total of 337 adverse events have been reported, from which 34 were classified as serious.
  The 337 reported events correspond to 277 different subjects. 83% of reported events are pertaining to one single patient, 13.4% of subjects have more than one adverse event, 3.2% have 3 reported events and one patient (0.4%) had 6 reported adverse events.
Groups:
- Paroxysmal and Persistent Atrial Fibrillation: Patients with paroxysmal or persistent AF who meet the criteria for the crioablation of the pulmonary veins. Events analyzed globally, no per groups.
Arm/Group | Paroxysmal and Persistent Atrial Fibrillation
All-Cause Mortality (participants affected / at risk) | 5/1742
Serious Adverse Events (participants affected / at risk) | 34/1742
Other Adverse Events (participants affected / at risk) | 262/1742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxysmal and Persistent Atrial Fibrillation (N=1742)
Adverse event related to procedure (Injury, poisoning and procedural complications) | 21 (21) — Temporal phrenic nerve palsy, access complications, Transient ST elevation
Adverse event related to AF not related to procedure (Cardiac disorders) | 12 (12) — cardiac arrhythmia, stroke,
Unexpected Serious Adverse Device Event (Infections and infestations) | 1 (1) — Non-ST elevation acute coronary syndrome, sepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxysmal and Persistent Atrial Fibrillation (N=1742)
Adverse event related to procedure (Injury, poisoning and procedural complications) | 95 (99)
Adverse event related to AF not related to procedure (Cardiac disorders) | 164 (201)
Unexpected Serious Adverse Device Event (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT02785991/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02785991/SAP_001.pdf